CLINICAL TRIAL: NCT06407414
Title: The Effect of Neuromuscular Exercise Program on Strength, Balance, Sleep Quality and Functionality in Patellofemoral Pain Syndrome
Brief Title: Effectiveness of Neuromuscular Exercise in Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar8
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (Active Comparator): classical physiotherapy methods
  Interventions: Other: control
- exercise (Experimental): In addition to classical physiotherapy methods, neuromuscular exercise protocol will be applied.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: control — classical physiotherapy methods
  Arms: control
Other: Exercise — In addition to classical physiotherapy methods, neuromuscular exercise protocol will be applied.
  Arms: exercise

SUMMARY:
The aim of the study is to investigate the effects of a neuromuscular exercise program on strength, balance, sleep quality and functionality in individuals with Patellofemoral pain syndrome.

DETAILED DESCRIPTION:
The research is planned as a quantitative study. Classical knee exercises will be given to 25 individuals in the control group of the study. An exercise program consisting of Neuromuscular exercises will be applied to 25 individuals in the intervention group. In data collection, strength and balance measurements will be measured face to face by a physiotherapist, and the scales to be made through a survey will be sent to the patients online and they will be asked to fill them out. The scales and forms to be used are as follows: 1.Kujala Patellofemoral Score Scale 2.Lysholm Knee Scoring Scale 3.International Physical Activity Survey 4.Pittsburgh Sleep Quality Index 5.Y Balance Test 6.30 Seconds Sit and Stand Test Applied scales will be done by the physiotherapist. The surveys will be uploaded to the Google Forms database and the participants will be contacted via e-mail or mobile phone applications (such as Whatsapp, Telegram) to participate. They will first be asked to fill out the surveys before starting the exercise program and they will be asked to apply the exercise program. It will be explained as follows. Exercises will be planned 3 times a week and for 12 weeks. Participants will be asked to participate in the survey again after completing the exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study.
* Not under 30 years of age and not over 60 years of age.
* Having patellofemoral pain syndrome.
* Not having a physical disability.
* Not having undergone any knee-related surgery.
* Having access to a computer/tablet/phone and the internet.

Exclusion Criteria:

* Not accepting the voluntary consent form.
* Being under 30 years of age and over 60 years of age.
* Having undergone any knee-related surgery.
* Having cognitive, mental or psychological problems.
* Having impaired vision or hearing.
* Having a physical condition that causes significant loss of function.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Kujala Patellofemoral Score Scale | 14 weeks
  Kujala patellofemoral scoring is a tool that allows functional evaluation of knee complaints related to the patellofemoral structure. Different scoring systems have been developed for knee-specific symptoms; however, only a few of these are focused on patellofemoral pain.The Kujala Patellofemoral Score Scale is graded on a scale of 0 to 100, with 100 being the highest possible score.
Lysholm Knee Scoring Scale | 14 weeks
  The Lysholm knee scoring scale is a global assessment tool that reflects overall functional outcome and physical activity level. The Lysholm scale is an 8-item questionnaire originally designed to assess knee function after knee ligament injuries. It was later confirmed for other knee conditions. Items evaluated according to the Lysholm scale include pain, type of support, instability, locking, swelling, limping, climbing stairs, and squatting. All items are scored to yield a score of 1, ranging from 0 to 100, with a higher Lysholm score indicating a lower level of symptoms and a higher level of functioning (91-100 = excellent, 84-90 = good, 65-83 = fair).
International Physical Activity Survey | 14 weeks
  Provides information on time spent walking, moderate and vigorous activities, and time spent sitting. Calculation of the total score of the short form includes the sum of the duration (minutes) and frequency (days) of walking, moderate-intensity activity, and vigorous activity. The energy required for activities is calculated with the metabolic equivalent(MET) -minute score. Standard metabolic equivalent (MET) values have been established for these activities.
Pittsburgh Sleep Quality Index | 14 weeks
  The pittsburgh Sleep Quality Index is a quantitative measure of sleep quality to define good and bad sleep. It includes 24 questions in total. The self-assessment questions include various items related to sleep quality. The total score is between 0-21. A high total score indicates poor sleep quality. The index does not indicate the presence of sleep disturbances or the prevalence of sleep disturbances. However, a pittsburgh Sleep Quality Index total score of five or more indicates poor sleep quality
Y Balance Test | 14 weeks
  Y balance test is a simple but reliable test used to measure dynamic balance. The Y balance test is a dynamic test performed in a one-legged stance that requires strength, flexibility, core control and proprioception. It has been used to evaluate physical performance, demonstrate functional symmetry, and identify athletes at higher risk for lower extremity injury. With the test complete and all performances recorded, the test administrator can then calculate the athlete's Y Balance Test performance scores using any of, or all of, the following three equations:
  Absolute reach distance (cm) = (Reach 1 + Reach 2 + Reach 3) / 3 Relative (normalised) reach distance (%) = Absolute reach distance / limb length * 100 Composite reach distance (%) = Sum of the 3 reach directions / 3 times the limb length * 100
30 Second Sit and Stand Test | 14 weeks
  It is a test that evaluates the patient's sitting and standing activity, lower extremity strength and dynamic balance. The number of times the patient sits and stands within 30 seconds gives the score of the test. For this test performed to determine leg strength; A straight-backed chair with a seating height of 43.18cm (12-in) and no armrests is used. The individual is asked to sit in the middle of the chair with his back upright, his feet on the ground, and his arms crossed in front of his chest (right hand on the left shoulder, left hand on the right shoulder). While in this position, the individual starts the test with the start command and takes off as fully as he can during 30 seconds. The number of complete starts he makes during 30 seconds constitutes the subject's score.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra ARISÜT, Study Chair — Uskudar University
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basbug P, Kilic RT, Atay AO, Bayrakci Tunay V. The effects of progressive neuromuscular exercise program and taping on muscle strength and pain in patellofemoral pain. A randomized controlled blind study. Somatosens Mot Res. 2022 Mar;39(1):39-45. doi: 10.1080/08990220.2021.1987877. Epub 2021 Oct 29. PMID 34713770
- [Background] Kim S, Roh Y, Glaviano NR, Park J. Quadriceps Neuromuscular Function During and After Exercise-Induced Fatigue in Patients With Patellofemoral Pain. J Athl Train. 2023 Jun 1;58(6):554-562. doi: 10.4085/1062-6050-0348.22. PMID 36395370
- [Background] Kolle T, Alt W, Wagner D. Effects of a 12-week home exercise therapy program on pain and neuromuscular activity in patients with patellofemoral pain syndrome. Arch Orthop Trauma Surg. 2020 Dec;140(12):1985-1992. doi: 10.1007/s00402-020-03543-y. Epub 2020 Jul 29. PMID 32728976
- [Background] Rathleff MS, Samani A, Olesen JL, Roos EM, Rasmussen S, Madeleine P. Effect of exercise therapy on neuromuscular activity and knee strength in female adolescents with patellofemoral pain-An ancillary analysis of a cluster randomized trial. Clin Biomech (Bristol). 2016 May;34:22-9. doi: 10.1016/j.clinbiomech.2016.03.002. Epub 2016 Mar 11. PMID 27054583
- [Background] Saltychev M, Dutton RA, Laimi K, Beaupre GS, Virolainen P, Fredericson M. Effectiveness of conservative treatment for patellofemoral pain syndrome: A systematic review and meta-analysis. J Rehabil Med. 2018 May 8;50(5):393-401. doi: 10.2340/16501977-2295. PMID 29392329